CLINICAL TRIAL: NCT02082184
Title: Randomised Controlled Study to Evaluate the Impact of Novel Glucose Sensing Technology on HbA1c in Type 2 Diabetes
Brief Title: An Evaluation of a Novel Glucose Sensing Technology in Type 2 Diabetes
Acronym: REPLACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADC-CI-APO-12018
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Sensing Technology; Type 2 Diabetes,
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensor Based Glucose Monitoring System (Experimental): Standard system use for 6 months. Followed by open access to the device for 6 months.
  Interventions: Device: Sensor Based Glucose Monitoring System
- Standard Blood Glucose Monitoring (Active Comparator): Subjects randomised to the control group will be given blood glucose meters for monitoring for the 6 months study duration.
  Interventions: Device: Standard Blood Glucose Monitoring

INTERVENTIONS:
Device: Sensor Based Glucose Monitoring System — Subjects will wear the Abbott Sensor Based Glucose Monitoring System (unmasked) for 6 months to monitor their glucose levels. Post completion of the 6 month intervention, subjects participating in this arm of the study will be given a further 6 month period of open access to the device.
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation.
  Arms: Sensor Based Glucose Monitoring System
Device: Standard Blood Glucose Monitoring — Subjects will use an Abbott Blood Glucose Monitoring System (standard blood glucose meter) for 6 months to monitor their glucose levels. A 14-day masked wear of the Abbott Sensor Based Glucose Monitoring System is included for these subjects at the 6 month time point, to collect glycaemic variability data for comparison to the intervention group of the study.
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation.
  Arms: Standard Blood Glucose Monitoring

SUMMARY:
To evaluate the impact of the Abbott Sensor Based Glucose Monitoring System on glycaemic control (HbA1c) compared to Self Monitoring Blood Glucose (SMBG) testing using a randomised controlled study design in adults with Type 2 diabetes using insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Has Type 2 diabetes on insulin therapy for ≥ 6 months and on their current regimen for ≥3 months prior to study entry.
2. Their insulin management must be one of the following;

   1. an injection regimen of prandial insulin at least once daily,
   2. or, prandial insulin at least once daily plus basal insulin at least once daily,
   3. or, continuous subcutaneous insulin infusion (CSII) with no plans to change during the study.
3. HbA1c result ≥7.5% (58 mmol/mol) and ≤12.0% (108 mmol/mol) on entry to the study.
4. Reports self-testing of blood glucose levels on a regular basis equivalent to a minimum of 10 tests per week, for at least 2 months prior to study entry.
5. In the investigator's opinion the subject is considered technically capable of using the Abbott Sensor Based Glucose Monitoring System.
6. In the Investigator's opinion the subject is proactive and therefore willing to modify their diabetes management
7. Aged 18 years or over.

Exclusion Criteria:

1. Insulin regimen consists entirely of basal or includes bi-phasic insulin.
2. Subject is currently prescribed animal insulin.
3. Subject is currently prescribed steroid therapy or is likely to require steroid therapy for any acute or chronic condition during the study.
4. Has known allergy to medical grade adhesives.
5. Currently participating in another device or drug study that could affect glucose measurements or glucose management.
6. Currently using a Continuous Glucose Monitoring (CGM) device or has used one within the previous 4 months.
7. Is planning to use a CGM device at any time during the study.
8. Total daily dose of insulin (TDD) is >1.75iu/kg at entry to the study.
9. A female subject who is pregnant or planning to become pregnant within the study duration.
10. Currently receiving dialysis treatment or planning to receive dialysis during the study.
11. Has experienced an acute myocardial infarction within previous 6 months.
12. Has a concomitant disease or condition that may compromise patient safety, including unstable coronary heart disease, cystic fibrosis, serious psychiatric disorder, or any other uncontrolled medical condition.
13. Has a pacemaker or any other neuro stimulators.
14. Has experienced any episode of severe hypoglycaemia, requiring third party assistance and/or admission to hospital, in the previous 6 months.
15. Has experienced any episode of diabetic ketoacidosis (DKA) or hyperosmolar hyperglycaemic state (HHS) in the previous 6 months.
16. In the investigator's opinion, the subject is considered as unsuitable for inclusion in the study for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Haak, Principal Investigator — Research Institute of Diabetes Academy Mergentheim (FIDAM)
Locations (26):
- France (8):
  - CHU Haut Lévêque, Bordeaux
  - Hôpital sainte Marguerite, Marseille
  - CHU Lapeyronie, Montpellier
  - CHU. Nancy, Nancy
  - Hopital Guillaume et René Laennec, Nantes
  - Hospital Lariboisere, Paris
  - Hôpital Cochin, Paris
  - Hôpital Rangueil, Toulouse
- Germany (10):
  - Diabetes Zentrum Mergentheim, Bad Mergentheim
  - Praris Dr Karin Schlecht, Eisenach
  - Diabetologische Schwenpunlet Praxis, Hamburg
  - Gemeiusilaftsproxis Fur Junere,, Hamburg
  - Vorstandsmitglied Deutsche Diabetes-Hilfe, Hamburg
  - Hohenzollernring, Münster
  - Diabetes Center Quakenbruck, Quakenbrück
  - Diabetes Schwerpunktpraxis Loccum, Rehburg-Loccum
  - An der Pforte, Rosenheim
  - Versdias GmbH, Sulzbach-Rosenberg
- United Kingdom (8):
  - Ayr Hospital, Ayr, Ayrshire
  - Diabetes Research, Linda McCartney Centre, Royal Liverpool University Hospital, Liverpool, Cheshire
  - Royal United Hospital, Bath
  - FRCPath Life and Health Sciences, Aston University, Birmingham
  - University Hospital of North Durham, Durham
  - The Diabetes Centre, Ipswich Hospital NHS Trust, Ipswich
  - St. James University Hospital, Leeds Teaching Hospitals NHS Trust, Leeds
  - Rotherham General Hospital, Rotherham

REFERENCES:
- [Derived] Rayman G, Kroger J, Bolinder J. Could FreeStyle Libre sensor glucose data support decisions for safe driving? Diabet Med. 2018 Apr;35(4):491-494. doi: 10.1111/dme.13515. Epub 2017 Oct 14. PMID 28945936
- [Derived] Haak T, Hanaire H, Ajjan R, Hermanns N, Riveline JP, Rayman G. Use of Flash Glucose-Sensing Technology for 12 months as a Replacement for Blood Glucose Monitoring in Insulin-treated Type 2 Diabetes. Diabetes Ther. 2017 Jun;8(3):573-586. doi: 10.1007/s13300-017-0255-6. Epub 2017 Apr 11. PMID 28401454
- [Derived] Haak T, Hanaire H, Ajjan R, Hermanns N, Riveline JP, Rayman G. Flash Glucose-Sensing Technology as a Replacement for Blood Glucose Monitoring for the Management of Insulin-Treated Type 2 Diabetes: a Multicenter, Open-Label Randomized Controlled Trial. Diabetes Ther. 2017 Feb;8(1):55-73. doi: 10.1007/s13300-016-0223-6. Epub 2016 Dec 20. PMID 28000140

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 302 subjects consented and enrolled into the study. Seventy-eight (78) of these failed screening or withdrew before randomisation. Two hundred and twenty-four (224) subjects were randomised and 201 completed the study.
Groups:
- Sensor Based Glucose Monitoring System: Standard system use for 6 months. Followed by open access to the device for 6 months.
  Sensor Based Glucose Monitoring System: Subjects will wear the Abbott Sensor Based Glucose Monitoring System (unmasked) for 6 months to monitor their glucose levels. Post completion of the 6 month intervention, subjects participating in this arm of the study will be given a further 6 month period of open access to the device.
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation.
- Standard Blood Glucose Monitoring: Subjects randomised to the control group will be given blood glucose meters for monitoring for the 6 months study duration.
  Standard Blood Glucose Monitoring: Subjects will use an Abbott Blood Glucose Monitoring System (standard blood glucose meter) for 6 months to monitor their glucose levels. A 14-day masked wear of the Abbott Sensor Based Glucose Monitoring System is included for these subjects at the 6 month time point, to collect glycaemic variability data for comparison to the intervention group of the study.
  All subjects will wear a masked Abbott Sensor Based Glucose Monitoring System, for 14 days prior to randomisation.
Period: Overall Study
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Started | 149 | 75
Completed | 139 | 62
Not Completed | 10 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Medical diagnosis | 1 | 2
Not completed — Device associated symptoms | 5 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 0 | 6
Not completed — Lost to Follow-up | 0 | 2
Not completed — Subject non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring | Total
Number analyzed (Participants) | 149 | 75 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.9) | 59.5 (11.0) | 59.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 19 | 74
  Male | 94 | 56 | 150
Screening HbA1c [Mean (Standard Deviation); unit: %] | 8.74 (0.97) | 8.88 (1.04) | 8.79 (0.99)
Screening HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 72.0 (10.6) | 73.5 (11.3) | 72.5 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c at 6 Months
Description: Difference in HbA1c between intervention and control group at day 194 adjusting for baseline HbA1c at day 1 using ANCOVA.
Time Frame: Baseline and Day 194
Measure: Mean (Standard Deviation); unit: percentage of Glycated Haemoglobin
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 149 | 75
percentage of Glycated Haemoglobin
  Baseline | 8.65 (1.01) | 8.75 (0.98)
  Day 194 | 8.37 (0.83) | 8.34 (1.14)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Test type: Superiority or Other; p = 0.8222, ANCOVA; Mean Difference (Final Values) = 0.03, Standard Error of Mean 0.114

2. Secondary Outcome: Time in Range
Description: Difference in time in range 70-180 mg/dL between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15 time in range) using ANCOVA.
Time Frame: Baseline and Days 194 to 208
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 149 | 75
hours per day
  Baseline | 13.9 (4.5) | 13.5 (5.2)
  Days 194-208 | 13.6 (4.6) | 13.2 (4.9)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Test type: Superiority or Other; p = 0.7925, ANCOVA; Mean Difference (Final Values) = 0.2, Standard Error of Mean 0.58

3. Secondary Outcome: Time Spent <70 mg/dL and <55 mg/dL
Description: Difference in time <70 mg/dL and <55 mg/dL (hours per day) between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15) using ANCOVA.
Time Frame: Baseline and Days 194 to 208
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 149 | 75
hours per day
  Time spent <70 mg/dL, Baseline | 1.30 (1.78) | 1.08 (1.58)
  Time spent <70 mg/dL, Days 194-208 | 0.59 (0.82) | 0.99 (1.29)
  Time spent <55 mg/dL, Baseline | 0.59 (1.13) | 0.38 (0.83)
  Time spent <55 mg/dL, Days 194-208 | 0.19 (0.37) | 0.37 (0.69)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of time spent <70 mg/dL; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.47, Standard Error of Mean 0.134
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of time spent <55 mg/dL; Test type: Superiority or Other; p = 0.0014, ANCOVA; Mean Difference (Final Values) = -0.22, Standard Error of Mean 0.068

4. Secondary Outcome: Frequency of Episodes <70 mg/dL and <55 mg/dL
Description: Difference in frequency of episodes <70 mg/dL and <55 mg/dL (number per day) between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15) using ANCOVA.
Time Frame: Baseline and Days 194 to 208
Measure: Mean (Standard Deviation); unit: number of episodes per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 149 | 75
number of episodes per day
  Frequency of episodes <70 mg/dL, Baseline | 0.64 (0.63) | 0.63 (0.66)
  Frequency of episodes <70 mg/dL, Days 194-208 | 0.38 (0.45) | 0.53 (0.59)
  Frequency of episodes <55 mg/dL, Baseline | 0.34 (0.50) | 0.27 (0.44)
  Frequency of episodes <55 mg/dL, Days 194-208 | 0.14 (0.24) | 0.24 (0.36)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of frequency of episodes <70 mg/dL; Test type: Superiority or Other; p = 0.0164, ANCOVA; Mean Difference (Final Values) = -0.16, Standard Error of Mean 0.065
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of frequency of episodes <55 mg/dL; Test type: Superiority or Other; p = 0.0017, ANCOVA; Mean Difference (Final Values) = -0.12, Standard Error of Mean 0.037

5. Secondary Outcome: Time Spent >180 mg/dL and >240 mg/dL
Description: Difference in time >180 mg/dL and >240mg/dL (hours per day) between intervention and control group assessed in days 194 to 208 adjusting for baseline (days 1 to 15) using ANCOVA.
Time Frame: Baseline and Days 194 to 208
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 149 | 75
hours per day
  Time spent >180 mg/dL, Baseline | 8.8 (5.0) | 9.4 (5.8)
  Time spent >180 mg/dL, Days 194-208 | 9.8 (4.8) | 9.8 (5.4)
  Time spent >240 mg/dL, Baseline | 3.1 (3.3) | 3.9 (4.5)
  Time spent >240 mg/dL, Days 194-208 | 3.5 (3.7) | 3.9 (4.2)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of time spent >180 mg/dL; Test type: Superiority or Other; p = 0.5970, ANCOVA; Mean Difference (Final Values) = 0.3, Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Statistical analysis of time spent >240 mg/dL; Test type: Superiority or Other; p = 0.8729, ANCOVA; Mean Difference (Final Values) = 0.1, Standard Error of Mean 0.46

6. Secondary Outcome: Number of Glucose Measurements Performed
Description: Number of blood glucose fingerstick tests per day by intervention and control group during days 15 to 208. The number of sensor scans performed by the intervention group during days 15 to 208.
Time Frame: Days 15 to 208
Measure: Mean (Standard Deviation); unit: number of measurements per day
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 132 | 52
number of measurements per day
  Number of fingerstick tests, Days 194-208 | 0.4 (1.0) | 3.8 (1.9)
  Number of sensor scans, Days 15-208 | 8.3 (4.4) | NA (NA) — Number of sensor scans does not apply to this group as they did not use the sensor.

7. Secondary Outcome: System Utilisation
Description: Sensor utilisation assessed by percentage of sensor glucose data collected by the intervention group.
Time Frame: Days 15 to 208
Population: 138 subjects included in the analysis, 11 were not included due to missing data.
Measure: Mean (Standard Deviation); unit: percentage of sensor glucose collected
Arm/Group | Sensor Based Glucose Monitoring System
Number analyzed (Participants) | 138
percentage of sensor glucose collected | 88.7 (9.2)

8. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQc) Scores From Day 1 to Day 194.
Description: The Diabetes Treatment Satisfaction Questionnaire change (DTSQc) score is used to assess relative change in participant satisfaction from baseline. The questionnaire consists of 8 items, 6 of which (1 and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale (which ranges from -3 (much less satisfied) to +3 (much more satisfied). The scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from -18 (much less satisfied) to +18 (much more satisfied).
  There is one question to assess the change in perceived frequency of Hypoglycaemia and one question to assess change in perceived frequency of Hyperglycaemia. Each question is rated on a 7-point Likert scale (-3 to +3), -3 (much less of the time now) to +3 (much more of the time now).
  The ANCOVA adjusts for baseline DTSQs (status version).
Time Frame: Baseline and Day 194
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Number analyzed (Participants) | 121 | 50
units on a scale
  Hyperglycaemia | 0.3 (1.9) | 0.2 (1.7)
  Hypoglycaemia | -0.2 (1.6) | 0.0 (1.4)
  Treatment Satisfaction | 13.4 (4.3) | 9.6 (5.6)
Statistical Analysis 1: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Perceived frequency of hyperglycaemia; Test type: Superiority or Other; p = 0.6075, ANCOVA; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Perceived frequency of hypoglycaemia; Test type: Superiority or Other; p = 0.2295, ANCOVA; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Sensor Based Glucose Monitoring System vs Standard Blood Glucose Monitoring; Total treatment satisfaction score; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.1, Standard Error of Mean 0.80

ADVERSE EVENTS:
Time Frame: Adverse events collected from enrolment (6 months)
Description: In addition to the serious adverse events listed below, 1 subject who withdrew from the study before randomisation reported serious adverse events of hypoglycaemia and renal impairment.
  No serious adverse events were related to the study device.
Arm/Group | Sensor Based Glucose Monitoring System | Standard Blood Glucose Monitoring
Serious Adverse Events (participants affected / at risk) | 16/149 | 12/75
Other Adverse Events (participants affected / at risk) | 49/149 | 27/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor Based Glucose Monitoring System (N=149) | Standard Blood Glucose Monitoring (N=75)
acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
cerebellar ischemia (Nervous system disorders) | 0 (0) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
chest pain (General disorders) | 1 (1) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
oesophagael carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
pancreatic neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
retinal detachment (Eye disorders) | 1 (1) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor Based Glucose Monitoring System (N=149) | Standard Blood Glucose Monitoring (N=75)
Nasopharyngitis (Infections and infestations) | 30 (32) | 10 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 6 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 10 (27) | 7 (30)
Low density lipoprotein increased (Investigations) | 3 (3) | 4 (4)
Blood cholesterol increased (Investigations) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days